CLINICAL TRIAL: NCT04434807
Title: Ultra-Early, Minimally inVAsive intraCerebral Haemorrhage evacUATion Versus Standard trEatment (EVACUATE)
Brief Title: Ultra-Early, Minimally inVAsive intraCerebral Haemorrhage evacUATion Versus Standard trEatment
Acronym: EVACUATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Bruce Campbell, Professorial Fellow, Department of Medicine, Royal Melbourne Hospital, Faculty of Medicine, Dentistry and Health Sciences, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBC2001
Record Dates: First submitted 2020-06-13; First posted 2020-06-17 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Intra Cerebral Hemorrhage; Stroke
Keywords: neurosurgery; minimally invasive
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Intervention Model Description: Patients will receive either minimally invasive hematoma evacuation or standard medical therapy
Who Masked: Outcomes Assessor
Masking Description: The primary outcome of Modified Rankin scale (mRS) and secondary outcomes including National Institutes of Health Stroke Scale (NIHSS) are assessed by a blinded clinician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Minimally invasive hematoma evacuation (Experimental): Patients randomized to minimally invasive hematoma evacuation will have neurosurgery followed by standard medical therapy in a stroke care unit or intensive care unit, as appropriate to the patients clinical condition.
  Interventions: Procedure: Minimally invasive hematoma evacuation
- Standard care (medical therapy) (No Intervention): Patients randomized to medical management will receive the standard medical therapies for the treatment of intracerebral hemorrhage in a stroke care unit or intensive care unit, as appropriate to the patients clinical condition, with no planned surgical intervention.

INTERVENTIONS:
Procedure: Minimally invasive hematoma evacuation — Neurosurgery performed via burr hole or minicraniotomy and using the Aurora surgiscope and evacuator (Integra Lifesciences)
  Arms: Minimally invasive hematoma evacuation

SUMMARY:
A randomized controlled trial of ultra-early, minimally invasive, hematoma evacuation versus standard care within 8 hours of intracerebral hemorrhage. Patients presenting to the emergency department with stroke due to supratentorial, spontaneous intracerebral hemorrhage >20mL volume will be assessed to determine their eligibility for randomization into the trial. If the patient gives informed consent they will be randomized 50:50 using central computerized allocation to minimally invasive hematoma evacuation using the Aurora surgiscope and evacuator (Integra Lifesciences) versus standard medical therapy. The trial is prospective, randomized, open-label, blinded endpoint (PROBE) design with seamless phase 2b-3 transition if the intermediate endpoint (successful hematoma evacuation) is met in analysis of the first 52 patients. Adaptive sample size re-estimation (Mehta and Pocock) will be performed when 160 patients have completed 6 month follow-up (minimum sample size 240, maximum sample size 434).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an acute supratentorial intracerebral hemorrhage (ICH) ≥20mL in volume
2. Age ≥18 years
3. Surgery can commence within 8 hours of symptom onset (the time the patient was last known to be well) or, in patients with wake-up onset, within 8 hours of the time the patient awoke with symptoms. Patients presenting with small ICH (volume <20mL) with clinical deterioration judged due to ICH hematoma expansion meeting volume criteria may be randomized if surgery can commence within 8 hours of clinical deterioration
4. Moderate neurological deficit (NIHSS≥6)
5. Pre-stroke mRS ≤3 (independent function or requiring only minor domestic assistance and able to manage alone for at least 1 week).
6. CTA or MRA is performed and does not show an underlying vascular lesion

Exclusion Criteria:

1. Brainstem ICH
2. ICH secondary to trauma, where brain injury is judged more likely to be due to the broad effects of trauma rather than the focal ICH.
3. Hereditary or acquired hemorrhagic diathesis or coagulation factor deficiency (in liver disease, INR>1.4).
4. Platelet count <75,000
5. Unreversible heparinization or anticoagulation. If reversing warfarin, INR should be ≤1.4 before procedure commences. Reversal of heparin by protamine, dabigatran by idarucizumab and rivaroxaban, apixaban and enoxaparin by andexanet (where available) is permitted. Unreversed anticoagulation with a last dose within 48 hours is an exclusion.
6. Recent (<12 hours) parenteral GPIIb/IIIa antagonist.
7. Recent (<1 hour) thrombolysis. If the ICH has occurred between 1 and 12 hours following thrombolysis, cryoprecipitate (1U per 10kg) and tranexamic acid must be administered prior to treatment.
8. Participation in any investigational study in the last 30 days
9. Pregnant women (clinically evident)
10. Co-morbidities or advance care directive preventing general anaesthesia for the procedure.
11. Known terminal illness such that the patients would not be expected to survive a year.
12. Planned withdrawal of care or comfort care measures.
13. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dichotomized Modified Rankin Scale Score 0-3 vs. 4-6 at 6 months post-onset (Adjusted) | 6 months post-stroke
  Modified Rankin Scale (mRS) 0-3 at 6 months, adjusted for age, baseline GCS, immediate pre-treatment ICH volume and immediate pre-treatment IVH volume.

SECONDARY OUTCOMES:
Dichotomized Modified Rankin Scale Score 0-2 or no change from baseline vs. 3-6 at 6 months post-onset (adjusted) | 6 months post-stroke
  Modified Rankin Scale (mRS) 0-2 or no change from baseline at 6 months, adjusted for age, baseline GCS, immediate pre-treatment ICH volume and immediate pre-treatment IVH volume
Ordinal analysis of Modified Rankin Scale Score at 6 months post-onset (adjusted) | 6 months post-stroke
  Ordinal analysis of Modified Rankin Scale Score (merging mRS 5-6) at 6 months, adjusted for age, baseline GCS, immediate pre-treatment ICH volume and immediate pre-treatment IVH volume
Utility-weighted analysis of Modified Rankin Scale Score at 6 months post-onset (adjusted) | 6 months post-stroke
  Utility-weighted analysis of Modified Rankin Scale Score at 6 months, adjusted for age, baseline GCS, immediate pre-treatment ICH volume and immediate pre-treatment IVH volume
Reduction in hematoma volume at 24 hours >70% or <15mL residual volume (adjusted) | 24 hours post-randomization
  Reduction in hematoma volume at 24 hours >70% or <15mL residual volume, adjusted for immediate pre-treatment ICH volume
Proportion of patients with early neurological improvement at 7 days (adjusted) | 7 days post-stroke
  Proportion of patients with ≥8 point reduction in National Institutes of Health Stroke Scale (NIHSS) score or reaching 0-1 at 7 days (or at discharge if earlier) adjusted for baseline NIHSS and age

OTHER OUTCOMES:
Safety: Death due to any cause at 6 months (adjusted) | 6 months post-stroke
  Death due to any cause at 6 months, adjusted for age, baseline GCS, immediate pre-treatment ICH volume and immediate pre-treatment IVH volume.
Safety: Hematoma growth or reaccumulation at 24 hours | 24 hours post-randomization
  Hematoma growth or reaccumulation defined as >33% or >6mL increased volume between baseline and 24 hour scans (or in the intervention arm a hematoma volume on the follow-up scan exceeding the immediate pre-treatment volume), adjusted for the pre-treatment ICH volume.
Intermediate outcome measure (primary outcome measure for Phase 2b component): Reduction in hematoma volume at 24 hours >70% or <15mL residual volume (adjusted) | 24 hours post-randomization
  Intermediate outcome measure (primary outcome measure for the Phase 2b component to be analysed for the first 52 patients): Reduction in hematoma volume at 24 hours >70% or <15mL residual volume, adjusted for immediate pre-treatment ICH volume
Patient Reported Outcomes Measurement Information System (PROMIS10) | 6 and 12 months post-stroke
Modified Rankin Scale (mRS) 0-2, 0-3, ordinal and utility-weighted analysis at 12 months | 12 months post-stroke
Assessment of Quality of Life (EQ5D) at 12 months | 12 months post-stroke
  Assessment of Quality of Life (EQ5D) at 12 months (mapped to mRS at baseline)
Length of stay in intensive care unit, acute hospital, acute hospital and rehabilitation | 6 months post-stroke
Home time - time spent at home in the first 6 months | 6 months post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kleinig, Principal Investigator — Royal Adelaide Hospital/University of Adelaide; Amal Abou-Hamden, Principal Investigator — Royal Adelaide Hospital/University of Adelaide; John Laidlaw, Principal Investigator — Royal Melbourne Hospital/University of Melbourne; J Mocco, Principal Investigator — Icahn School of Medicine, Mt Sinai Hospital, New York; Christopher Kellner, Principal Investigator — Icahn School of Medicine, Mt Sinai Hospital, New York; Stephen Davis, Principal Investigator — Royal Melbourne Hospital/University of Melbourne; Bruce Campbell, Principal Investigator — Royal Melbourne Hospital/University of Melbourne
Locations (13):
- Australia (13):
  - John Hunter Hospital, Newcastle, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - The Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - The Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - The Austin Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient data will be uploaded to the Virtual Stroke Trials Archive (http://www.virtualtrialsarchives.org/vista/) 2 years after the publication of the primary manuscript. Qualified investigators can access data after submission of a project proposal that has been approved by the VISTA-ICH steering committee.
Time Frame: 2 years after the publication of the primary manuscript
Access Criteria: Qualified investigators can access data after submission of a project proposal that has been approved by the VISTA-ICH steering committee.